CLINICAL TRIAL: NCT05136807
Title: Quality of Life in Patients With Asymptomatic Monoclonal Gammopathies
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-0172; NCI-2021-11118 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0172 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-11-11; First posted 2021-11-29 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Monoclonal Gammopathy of Undetermined Significance; Smoldering Plasma Cell Myeloma
MeSH Terms: conditions — Monoclonal Gammopathy of Undetermined Significance; Smoldering Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (quality of life questionnaire): Patients complete quality of life questionnaires over 10-15 minutes at baseline and every 6 months for patients participating in an observational study or every month for patients participating in a treatment study for up to 3 years.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Other: Quality-of-Life Assessment — Complete questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study examines the quality of life in patients with monoclonal gammopathy of unknown significance and smoldering multiple myeloma. Collecting quality of life information from patients may help doctors learn more about the most common symptoms and concerns patients with monoclonal gammopathy of unknown significance and smoldering multiple myeloma may have.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Describe baseline and follow up quality of life and monoclonal gammopathy of unknown significance/smoldering multiple myeloma (MGUS/SMM) related anxiety of patients with MGUS/SMM already participating in clinical trials at MD Anderson Cancer Center.

SECONDARY OBJECTIVE:

I. Identify the most common symptoms/patients concerns to evaluate future interventions for treatment/prevention in this population.

OUTLINE:

Patients complete quality of life questionnaires over 10-15 minutes at baseline and every 6 months for patients participating in an observational study or every month for patients participating in a treatment study for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either monoclonal gammopathy of unknown significance age >= 18 years old.

  * Both criteria must be met:

    * Serum monoclonal protein < 3 g/dL or urinary monoclonal protein < 500 mg per 24 hours and clonal bone marrow plasma cells < 10%
    * Absence of myeloma defining events or amyloidosis
* OR Patients with smoldering multiple myeloma age >= 18 years old.

  * Both criteria must be met:

    * Serum monoclonal protein >= 3 g/dL or urinary monoclonal protein >= 500 mg per 24 hours and/or clonal bone marrow plasma cells 10-60%
    * Absence of myeloma defining events or amyloidosis
* Patients must be enrolled in clinical trials for SMM or MGUS at MD Anderson Cancer Center, including protocols PA15-0575 (NCT02726750) (Prospective observational study of clinical and genomic predictors of progression to myeloma in asymptomatic monoclonal gammopathies); 2015-0148 (Phase II single arm trial of Isatuximab in patients with intermediate and high risk smoldering multiple myeloma); and 2015-0371 (NCT02603887) (Pilot single arm, single center, open label trial of Pembrolizumab in patients with intermediate and high risk smoldering multiple myeloma) and any future clinical trials for MGUS and/or SMM that open at MD Anderson Cancer Center.
* Only patients who are English or Spanish speaking are eligible.

Exclusion Criteria:

* Evidence of myeloma defining events or biomarkers of malignancy due to underlying plasma cell proliferative disorder meeting at least one of the following

  * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than the upper limit of normal or > 2.75 mmol/L (> 11 mg/dL)
  * Renal Insufficiency: creatinine clearance < 40 ml/min or serum creatinine > 2 mg/dL
  * Anemia: hemoglobin value < 10 g/dL or 2 g/dL < normal reference
  * Bone lesions: one or more osteolytic lesions on skeletal radiography, computerized tomography (CT) or 2-deoxy-2[F-18] fluoro-D-glucose positron emission tomography CT (PET-CT).
  * Clonal bone marrow plasma cell percentage >= 60%
  * Involved: uninvolved serum free light chain ratio >= 100 measured by Freelite assay (The Binding Site Group, Birmingham, United Kingdom [UK])
  * >1 focal lesions on magnetic resonance imaging (MRI) studies, if the patient has an MRI done per eligibility criteria (each focal lesion must be 5 mm or more in size)
* Plasma cell leukemia.
* Presence of cognitive impairment or delirium as determined by the primary clinician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with monoclonal gammopathy of unknown significance or smoldering multiple myeloma at MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2016-06-07 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Quality of life questionnaires | Up to 3 years
  Patients complete quality of life questionnaires over 10-15 minutes at baseline.
  Score scale ranges from (1-4) 1 - Not at all and 4 - Almost all the time
Quality of life questionnaires | Up to 3 years
  Patients complete quality of life questionnaires every 6 months for patients participating in an observational study or every month for patients participating in a treatment study for up to 3 years.
  Score scale ranges from (1-4) 1 - Not at all and 4 - Almost all the time

CONTACTS AND LOCATIONS:
Overall Officials: Melody E Becnel, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org